CLINICAL TRIAL: NCT03816813
Title: Detection of Hepcidin in Saliva and Its Utility as a Diagnostic Marker for Iron Deficiency
Brief Title: Assessement of Hepcidin in Saliva in Human Volunteers
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Diego Moretti, PhD, Senior Scientist, Swiss Federal Institute of Technology
Other Study IDs: HepSa
Record Dates: First submitted 2019-01-21; First posted 2019-01-25 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-01

CONDITIONS: Hepcidin, Saliva
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood and saliva sampling — blood and saliva sampling

SUMMARY:
Iron deficiency with or without anemia is considered the most widespread nutritional deficiency in the world. To diagnose iron deficiency anemia (hemoglobin and ferritin measurement), a venous blood sample is necessary. Whole saliva is a potentially attractive fluid for disease biomarker discovery and diagnostic efforts, because it is readily available from most individuals, can be easily collected and the collection procedure is non-invasive. The iron storage protein ferritin is too big, to be secreted into saliva. However, the main iron regulatory protein hepcidin is a very small protein and there is some evidence for hepcidin detection in saliva. The production of serum hepcidin positively correlates with serum ferritin, thereby reflecting patient's iron status. Whether hepcidin is detectable in saliva and whether saliva hepcidin correlates with serum hepcidin with current assays, needs to be tested.

ELIGIBILITY:
Inclusion Criteria:

* Normal-weight (BMI 18-24.9kg/m2)
* fasting
* Participants Need to have brushed their teeth at least 1 hour before the visit

Exclusion Criteria:

* acute, chronic illness
* use of long-term medication other than contraception
* medical Problems known to affect Fe homeostasis
* smoking

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: healthy volunteers, male and female
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Saliva hepcidin | Day 1am
Serum hepcidin | Day 1am
Serum ferritin | Day 1am
  Iron Status parameter

SECONDARY OUTCOMES:
Hemoglobin | Day 1am
Transferrin receptor | Day 1am
  Iron Status parameter
c-reactive protein | Day 1am
  Inflammation parameter
alpha-glycoprotein | Day 1am
  Inflammation parameter
Saliva hepcidin | Day 1pm
  to assess variability in saliva hepcidin during the day
Saliva hepcidin | Day 2am
  to assess variability in saliva hepcidin in two samples measured at the same time of the day

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Human Nutrition, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No